CLINICAL TRIAL: NCT06664060
Title: Efficacy of Two Nutritional Supplements on Healing and Bone Density in the Jaws
Brief Title: Osteoimplant and Bone Healing
Acronym: Osteocic
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Francisco Javier Manzano-Moreno, PhD, DDS, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4042/CEIH/2024
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dimensional Changes; Bone Density
Keywords: vitamin d; vitamin c; bone density; dimensional changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteoimplant (Experimental)
  Interventions: Drug: osteoimplant
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: osteoimplant — 30 lower third molars will be selected and prescribed preoperative treatment with two units of Osteoimplant Complex® 5 days prior to surgery and postoperative treatment with one unit of Osteoimplant® for 8 weeks from the time of surgery. Both nutritional supplements will be administered every 24 hours.
  Arms: osteoimplant
Drug: Placebo — 30 lower wisdom teeth will be selected and prescribed placebo, both preoperatively 5 days prior to surgery and postoperatively for 8 weeks from the time of surgery.
  Arms: placebo

SUMMARY:
In view of the above and the possible improvements in terms of postoperative morbidity and tissue repair in oral surgery, this study is justified, the general objective of which would be:

'To evaluate the efficacy of perioperative oral administration of two nutritional supplements based on vitamins and antioxidants (Osteoimplant Complex® and Osteoimplant®), using mandibular third molar surgery as a study model, assessing postoperative symptomatology and bone density'.

The null hypothesis of this study is: 1) the administration of the perioperative nutritional complex (Osteoimplant Complex® and Osteoimplant®) did not improve postoperative symptoms and 2) neither did it increase bone density after lower third molar extraction.

DETAILED DESCRIPTION:
In view of the above and the possible improvements in terms of postoperative morbidity and tissue repair in oral surgery, this study is justified, the general objective of which would be:

'To evaluate the efficacy of perioperative oral administration of two nutritional supplements based on vitamins and antioxidants (Osteoimplant Complex® and Osteoimplant®), using mandibular third molar surgery as a study model, assessing postoperative symptomatology and bone density'.

The null hypothesis of this study is: 1) the administration of the perioperative nutritional complex (Osteoimplant Complex® and Osteoimplant®) did not improve postoperative symptoms and 2) neither did it increase bone density after lower third molar extraction.

Study design. It is a randomised clinical trial (RCT), double blind controlled (neither the patient nor the examiner collecting the data knows the allocation group) and split-mouth to evaluate the efficacy of the perioperative oral administration of two nutritional complexes on postoperative symptoms, wound healing and bone density 8 weeks after the extraction of a mandibular third molar.

Composition of the nutritional supplements. A. Preoperative nutritional supplement, Osteoimplant Complex®: Ovocet®, vitamin C 48.5mg, coenzyme Q10 41.3mg, zinc 35mg, beta carotene 10% 25mg, bioflavonoids citrus 60% 20.83mg, vitamin E, magnesium 15mg.

B. Postoperative nutritional supplement, Osteoimplant®: Ovocet®, collagen 350mg, calcium 300mg, vitamin D3 100 IU/mg, magnesium 8mg.

Target population:

All patients with two lower third molars in need of extraction.

Study or accessible population:

All patients attending the Master's Degree in Oral Surgery and Implantology of the University of Granada who present with two lower third molars in need of extraction.

All patients, after inclusion in the study, will undergo a clinical history and subsequent clinical examination. The clinical history will consist of an anamnesis, where the patient's personal details will be collected (name, age, sex, profession, address and telephone number), as well as family history, illnesses suffered, previous surgical interventions, drug allergies and current treatment. Subsequently, a physical examination will be carried out, consisting of inspection and palpation of the buccofacial territory.

To complement our examination and make a correct diagnosis, all patients will undergo a radiological study as a step prior to surgery, which will always consist of an orthopantomography and a CBCT in order to assess three-dimensionally the relationship with adjacent anatomical structures, which will also help us to have a prior measurement of the patient's bone density.

Once the diagnosis has been correctly made, the patient will be informed, both orally and in writing, of the possible complications that may arise in this type of surgery.

In the same way, if the inclusion criteria established for this study are met, each patient will be offered the possibility of participating in the study, explaining in detail the main objective, the surgical procedure and the different phases of treatment; all detailed in an information sheet that will be handed out for reading. In the case of acceptance to participate, all patients will sign the study-specific informed consent form.

For the sample size, a total of 60 lower third molars and 30 patients will be collected. The sample will be divided into 2 groups of 30 lower third molars each and randomised using a randomisation table.

Group A: 30 lower third molars will be selected and prescribed preoperative treatment with two units of Osteoimplant Complex® 5 days prior to surgery and postoperative treatment with one unit of Osteoimplant® for 8 weeks from the time of surgery. Both nutritional supplements will be administered every 24 hours.

Group B: 30 lower wisdom teeth will be selected and prescribed placebo, both preoperatively 5 days prior to surgery and postoperatively for 8 weeks from the time of surgery.

Pre-operative medication and nutritional supplementation:

* If belonging to the control group: placebo, 2/24 hours, 5 days prior to surgery.
* If test group : Osteoimplant Complex®, 2/24 hours, 5 days prior to surgery.

Postoperative medication and nutritional supplementation:

* If in control group: placebo, 1/24 hours, for 8 weeks.
* If test group : Osteoimplant®, 1/24 hours, for 8 weeks.
* Antibiotic treatment: amoxicillin 750 mg, 1/8 hours, for 5 days. In case of penicillin allergy, the drug of choice is clindamycin 300 mg 1/8 hours for 5 days.
* Analgesic and anti-inflammatory treatment: ibuprofen 400 mg 1/8 hours for 2 days, from the third day on demand. As rescue medication, paracetamol 1 g.

PRIMARY VARIABLE

1. Bone density and dimensional changes:

Bone density and dimensional changes shall be assessed by a surgeon previously instructed by a specialised radiologist, by means of CBCT scans performed before (T0) and 8 weeks after (T1) extraction to obtain thus:

1. dimensional changes, evaluating the horizontal and vertical dimensions of hard tissue taking as a reference the amelocentric limit (LAC) of the adjacent tooth, so as to assess whether there has been loss of hard tissue following extraction and healing. For this purpose, three sections (A, B and C) shall be made at 5, 7 and 9 mm, taking as point 0 the imaginary horizontal line marked by the LAC of the adjacent tooth.
2. Bone density obtained after 8 weeks of healing: it shall be evaluated by making axial cuts in sections A, B and C in such a way that an area of 3 mm2 is determined (this area shall be located at a fixed horizontal distance from the LAC of the anterior tooth to be determined in each case at the level of the furca of the tooth to be extracted). The average bone density (Hounsfield value) in each of these areas shall be calculated in order to calculate the average bone density of healing for each alveolus. Changes in bone density will be assessed by analysing the differences between T1 and T0.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting both lower third molars.
* Adult patients between 18 and 40 years of age.
* Anaesthetic risk ASA I-II (American Society of Anaesthesiologists classification) [14].
* Absence of drug or food allergies that could compromise our study (e.g. egg).
* Signed informed consent.

Exclusion Criteria:

* Age not between 18-40 years.
* Pregnant or breastfeeding women.
* Presenting decompensated metabolic disease.
* Poor periodontal status (≥10% plaque index and bleeding index).
* Patients who have undergone radiotherapy in the last five years.
* Patients who will not comply with the study guidelines.
* Unsigned informed consent.
* History of allergy to any study medication or related drugs (e.g. egg).
* Patients with a history of renal colic.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
diensional changes | From the extraction (T0) to 8 weeks after (T1) extraction
  Dimensional changes shall be assessed by a surgeon previously instructed by a specialised radiologist, by means of CBCT scans performed before (T0) and 8 weeks after (T1) extraction to obtain thus:
  Dimensional changes, evaluating the horizontal and vertical dimensions of hard tissue taking as a reference the amelocentric limit (LAC) of the adjacent tooth, so as to assess whether there has been loss of hard tissue following extraction and healing. For this purpose, three sections (A, B and C) shall be made at 5, 7 and 9 mm, taking as point 0 the imaginary horizontal line marked by the LAC of the adjacent tooth.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pisalsitsakul N, Pinnoi C, Sutanthavibul N, Kamolratanakul P. Taking 200 mg Vitamin C Three Times per Day Improved Extraction Socket Wound Healing Parameters: A Randomized Clinical Trial. Int J Dent. 2022 Mar 10;2022:6437200. doi: 10.1155/2022/6437200. eCollection 2022. PMID 35310461
- [Result] Olmedo-Gaya MV, Manzano-Moreno FJ, Munoz-Lopez JL, Vallecillo-Capilla MF, Reyes-Botella C. Double-blind, randomized controlled clinical trial on analgesic efficacy of local anesthetics articaine and bupivacaine after impacted third molar extraction. Clin Oral Investig. 2018 Dec;22(9):2981-2988. doi: 10.1007/s00784-018-2386-1. Epub 2018 Feb 15. PMID 29450738
- [Result] Insua A, Galindo-Moreno P, Miron RJ, Wang HL, Monje A. Emerging factors affecting peri-implant bone metabolism. Periodontol 2000. 2024 Feb;94(1):27-78. doi: 10.1111/prd.12532. Epub 2023 Oct 30. PMID 37904311